CLINICAL TRIAL: NCT03585569
Title: A Prospective, Open Label, Single Center Study of Patients With Multiple Sclerosis With Lower Extremity Spasticity Who Are Treated With Dysport
Brief Title: " Treating MS Patients With Lower Extremity Spasticity Using Dysport"
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neurology Center of New England P.C. (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAIRB-17-0093
Record Dates: First submitted 2018-03-16; First posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Multiple Sclerosis; Spasticity, Muscle
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity | interventions — abobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Biological: Abobotulinumtoxin A — Treating Patients with Multiple Sclerosis with lower extremity spasticity using Dysport (Abobotulinumtoxin A)
  Other Names: Dysport

SUMMARY:
The purpose of this study is to determine whether Dysport® (abobotulinumtoxinA) injections for lower extremity spasticity showed a significant reduction of lower extremity spasticity after being injected with Dysport® (abobotulinumtoxinA) in patients with MS.

DETAILED DESCRIPTION:
Primary Objective To evaluate the effect of Dysport® (abobotulinumtoxin A) on lower extremity spasticity (soleus, gastrocnemius, lateral gastrocnemius, medial gastrocnemius, flexor digitorum longus, flexor halluces longus, rectus femorus, vastus lateralis, lateral hamstrings, medial hamstrings, adductor magnus, adductor longus, adductor brevis, triceps surae, tibialis posterior or anterior tibialis).

Other Objectives

* To explore the effect of Dysport® on improvement in walking ability in patients with MS
* To explore the effect of Dysport® on quality of (QoL) in patients with MS. Primary Endpoint Absolute change from baseline in Modified Ashworth Scale (MAS) through 20 weeks of treatment.

Other Endpoints

* Change from baseline in MAS scores at Weeks 12, 16, and 20.
* Change from baseline on QoL based on patient reported outcome (PRO) measures on the MSWS-12, MSIS 29, pain scales (0-10 pain scale) the MSSS-88, and the Penn spasm frequency scale through 20 weeks of treatment.
* Change from baseline on the time 25 foot walk (T25FW) test with timed up and go (TUG) through 20 weeks of treatment.
* Change from baseline on expanded disability status scale (EDSS) score at Weeks 12, 16, 20.
* Change from baseline in speed, cadence, general symmetry, propulsion, stride length, T25FW, TUG using GWALK device for gait assessments through 20 weeks.
* Adverse events over 20 weeks
* Serious adverse events over 20 weeks

ELIGIBILITY:
Inclusion Criteria:Subjects who meet all of the following inclusion criteria will be eligible:

1. Male or female with confirmed diagnosis of MS1 over 18 years of age.
2. Patients with a clinically definite diagnosis of MS including patients with relapsing-remitting MS, primary progressive MS, progressive relapsing MS, and secondary progressive MS based on clinical history, physical exam, current or previous brain or spine MRI, CSF analysis will be used to specify the class of MS of the patient.
3. Patients with no prior exposure to any commercial Botulinum toxin or patients that have had previous exposure to commercial Botulimun toxin no less than four months after last injection.
4. Naïve patients having a MAS score ≥1 at baseline in any of the following muscles soleus, gastrocnemius, lateral gastrocnemius, medial gastrocnemius, flexor digitorum longus, flexor halluces longus, rectus femorus, vastus lateralis, lateral hamstrings, medial hamstrings, adductor magnus, adductor longus, adductor brevis.
5. Patients with prior exposure to commercial Botulinum having a MAS ≥1 at baseline in any of the following US Dysport label muscles such as the soleus, gastrocnemius, lateral gastrocnemius, medial gastrocnemius, flexor digitorum longus, flexor halluces longus, or muscles beyond the label such as the rectus femorus, vastus lateralis, lateral hamstrings, medial hamstrings, adductor magnus, adductor longus, adductor brevis, tibialis posterior EDSS score less than 7.0.
6. Penn spasm frequency scale at baseline greater than 2.
7. Functional outcomes such as walking speed T25FW baseline walking speed greater than 0.8.
8. Subjects that have agreed to participate and have signed an informed consent form.

   -

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria will not be eligible:

  1. Subjects having experienced a relapse within the previous 30 days.
  2. Recently initiated treatment on antispasmodic therapy or Ampyra within 30 days of screening.
  3. Subjects that have not maintained a steady dose of baclofen or other antispasmodics in the previous 30 days will be excluded.
  4. Pregnant or women who intend to become pregnant or breastfeeding women. Women of child bearing potential are required to use oral contraceptives, condoms, intrauterine device (IUD) diaphragm, spermicide, sexual abstinence or vasectomized partner. Female patients using contraception should continue to use contraception 3- 4 months post injection. Women of childbearing potential are defined as any female who has experienced menarche and who is NOT permanently sterile or postmenopausal. Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Using Dysport to treat lower extremity spasticty in patients diagnosed with Multiple Sclerosis. Improved walking ability and quality of life in 28 patients based on quality of life assessments and patient reported outcomes. | 20 weeks
  Using Dysport® (abobotulinumtoxin A) to treat patients diagnosed with Multiple Sclerosis with lower extremity spasticity .

SECONDARY OUTCOMES:
Mean change from baseline in Modified Ashworth Scale (MAS) | Baseline week 12, week 16, and week 20
  Mean change from baseline in Modified Ashworth Scale (MAS).. The Modified Ashworth Scale issued to grade spasticity. This scale measures the presence of velocity-dependent resistance on a 0 to 4 scale, with zero representing normal muscle tone, and four representing a limb that is fixed in flexion or extension

OTHER OUTCOMES:
12 item Multiple Sclerosis Walking scale (MSWS-12) Improvement | Baseline weeks 12, 16, and 20
  Mean change from baseline in the 12 Item Multiple Sclerosis Walking Scale. The Multiple Sclerosis Walking Scale is a self-assessment scale which measures the impact of MS on walking. It consists of 12 questions concerning the limitations to walking due to MS during the past 2 weeks. Each item can be answered with 5 options, with 1 meaning no limitation and 5 extreme limitation.
  A total score can be generated and transformed to a 0 to 100 scale by subtracting the minimum score possible (12) from the patient's score, dividing by the maximum score possible minus the minimum possible (60-12 or 48), and multiplying the result by 100. Walking improvement on the MSWS-12 is indicated by negative change scores
Improvement of (MSIS-29) Multiple Sclerosis Impact Scale | Baseline weeks 12,16 and 20
  Mean change from baseline in the (MISIS-29) Multiple Sclerosis Impact Scale.The MSIS-29 is a 29 item measurement, which assesses the physical and psychological impact of MS on affected individuals; it is a self report questionnaire consisting of 20 and 9 items, respectively. Scores on the individual items are added and then transformed to a 0-100 scale, thereby generating two summary scores (for physical and psychological impact). Higher scores indicate worse health.
Improvement of Pain Scale | Baseline weeks 12,16 and 20
  Mean change from baseline in the 0-10 Pain Scale. involves asking the patient to rate his or her pain from 0 to 10 (11 point scale) with the understanding that 0 is equal to no pain and 10 is equal to worst possible pain.
  0 Pain free
  1. Very minor annoyance-occasional minor twinges
  2. Minor annoyance-occasional
  3. Annoying enough to be distracting
  4. Can be ignored if you are really involved in your work, but still distracting,
  5. Can't be ignored for more than 30 minutes.
  6. Can't be ignored for any length of time, but you can still go to work and participate in social activities.
  7. Make it difficult to concentrate, interferes with sleep, you can still function with effort
  8. Physical activity severely limited. You can read and converse with effort. Nausea and dizziness may occur.
  9. Unable to speak, crying out or moaning uncontrollable- pain makes you pass out
  10. Unconscious. Pain makes you pass out.
Improvement of (MSSS-88) Multiple Sclerosis Spasticity Scale | Baseline weeks 12,16 and 20
  Mean Change from baseline in the (MSSS-88) Multiple sclerosis Spasticity scale measures patient experience and perception of the impact of spasticity in MS with day-to-day symptoms andduring functional activities over the previous two weeks. It has 88 questions to quantify spasticity for a total score and in eight clinically relevant and stand-alone subscales: muscle stiffness, pain and discomfort,muscle spasms, activities of daily living,walking, body movements, emotional health, and social functioning.This scale has 88 items that are rated on a 4-point scale of 1 (Not at all bothered) through 4 (Extremely bothered).
Improvement of the Penn Spasm frequency scale | Baseline weeks 12,16 and 20
  Mean change from baseline in the Penn Spasm frequency scale. The patient evaluates his/her "spasms", quantifying them according to 5 classifications (from 0 to 4).For ratings of 1 or greater, the severity of the spasms is also be evaluated, using a 3 level scale (mild, moderate or severe)
Improvement from baseline on the Timed 25 foot walk (T25FW) | Baseline weeks 12,16 and 20
  Mean change from baseline on the Timed 25 foot walk (T25FW) The Timed 25-Foot Walk test is a mobility and function test based on a timed 25-foot walk. An individual will be asked to walk 25 feet on a clearly marked course as quickly and safely as they can.
  The time is calculated with a stopwatch, recorded, and the individual is asked to repeat the task immediately, walking back the same distance to the their initial starting point.
Improvement of Timed up and Go | Baseline weeks 12,16 and 20
  Mean change from baseline on the Timed up and go. The purpose of the Timed Up and Go test is to identify individuals who are at risk of falling. It can screen for balance and gait problems.
  A person is observed as they stand from a sitting position without using their arms for support, then walk 10 feet, turn and return to a chair. Finally, they sit back in the chair without using their arms for support.
Improvement on the (EDSS) score | Baseline weeks 12,16 and 20
  Mean change from baseline on the Expanded Disability Status Scale (EDSS) score. is a 20 point ordinal scale ranging from 0 (normal neurological exam) to 10 (dead from MS). From 0-4.0, EDSS is determined by the combination of scores on 7 functional systems. From 4.0-6.0 EDSS is determined by the ability to walk a distance. EDSS 6.0 is the need for unilateral walking assistance. EDSS 6.5 is the need for bilateral walking assistance. Nonambulatory patients are scored EDSS ≥7.0, with higher number reflecting increasing difficulty with mobility and ability to perform self-care.
Walking improvement | Baseline weeks 12,16 and week 20
  Change from baseline in speed, cadence, general symmetry, propulsion, stride length using the G-Walk device is a wireless system of inertial sensors composed of a triaxial accelerometer, a magnetic sensor, and a triaxial gyroscope that, when positioned on L5 vertebrae of the spine, it allows for a functional objective gait analysis to be performed. The system extrapolates the data and calculates all the spatial-temporal gait parameters required to perform an assessment or to define a training strategy

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Q Napoli, MD, Principal Investigator — Neurology Center of New England P.C.
Locations (1):
- Neurology Center of New England P.C., Foxborough, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Poster and Paper with at AAN and ECTRIMS intention for full manuscript